CLINICAL TRIAL: NCT00766649
Title: Pilot Study of the Evaluation of Subconjunctival Sirolimus in the Treatment of Bilateral Geographic Atrophy Associated With Age-Related Macular Degeneration
Brief Title: Pilot Study of the Evaluation of Subconjunctival Sirolimus in the Treatment of Bilateral GA Associated With AMD
Acronym: SIRGA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090008; 09-EI-0008 (Registry Identifier: National Institutes of Health Clinical Center)
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Results first posted 2013-07-01 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2014-04

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age Related Macular Degeneration (AMD); Geographic Atrophy; Sirolimus; Age-Related Macular Degeneration; AMD
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus (Experimental): Participants receive a 20 μL (440 μg) subconjunctival injection of sirolimus in the study eye at baseline and every three months thereafter.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Participants receive a 20 μL (440 μg) subconjunctival injection of sirolimus in the study eye at baseline and every three months thereafter.
  Other Names: Rapamune®; rapamycin

SUMMARY:
This study will determine if a drug called sirolimus is safe to give to people with geographic atrophy GA and if it can help preserve vision in patients. GA is an advanced form of dry age-related macular degeneration (AMD). AMD affects the macula, the central part of the retina needed for sharp, clear vision. There are two types of AMD, wet and dry. In dry AMD, cells in the macula die.GA may at least partly be caused by inflammation. Sirolimus helps prevent inflammation and therefore may help treat GA.

People with GA in both eyes with visual acuity between 20/20 and 20/400 in each eye may be eligible for this study. Participants undergo the following tests and procedures:

* Sirolimus injections in the study eye at each 3-month clinic visit. The drug is injected under the outer layer of the eye after the patient receives antiseptic and numbing drops. Antibiotic drops are continued for 2 days after the injection.
* Eye examinations before the first injection, 1 month after the first injection, during each clinic visit (11 to 15 visits over 2 to 3 years) and 3 months after the final injection. The examination includes testing visual acuity, measuring eye pressure and checking eye movements. To examine the inside of the eye, the pupil is dilated with eye drops. Regular photographs of the inside of the eye and optical coherence tomography photographs, which allow measurement of the thickness of the retina, may be taken during the eye examination.
* Autofluorescence imaging. The patient sits in a chair with his or her head placed in a chin rest in front of a camera. A light in the camera is used to scan the eye.
* Blood tests. Blood is drawn at the first visit and at up to seven study visits to check blood chemistries, such as liver and kidney function.
* Urine pregnancy test for women who are able to become pregnant.

DETAILED DESCRIPTION:
Objective: Age-related macular degeneration (AMD), the leading cause of blindness in people over age 55 in the United States, is a heterogeneous clinical entity in which retinal degeneration occurs predominantly in the macula in the context of aging and leads to impairment of central visual acuity. AMD occurs in two general forms, one of which involves choroidal neovascularization (CNV) with subsequent formation of a disciform scar. This is often referred to as the neovascular or "wet" form. A second form, the subject of this study, is termed "dry" or atrophic macular degeneration and involves a constellation of clinical features that can include drusen, pigment clumping and/or retinal pigment epithelium (RPE) dropout and geographic atrophy (GA). GA can begin as a thinning of the RPE with involvement of the underlying choriocapillaris and lead subsequently to an atrophic change in the macula. Inflammation may play a role in the pathogenesis of GA. Sirolimus inhibits the production, signaling and activity of many inflammatory factors relevant to the development of GA. Therefore, the objective of this study is to investigate the safety and possible efficacy of multiple sirolimus subconjunctival injections in participants with bilateral GA.

Study Population: Ten participants with bilateral GA associated with AMD, with the potential to replace up to five participants if some fail to reach one year of follow-up.

Design: In this controlled, unmasked, Phase I/II study, one eye of eligible participants will be randomized to treatment while the fellow eye will be observed. Participants will receive a 20 μL (440 μg) subconjunctival injection of sirolimus in the study eye at baseline and every three months thereafter. The study will be completed once all participants have received two years of study medication and follow-up.

Outcome Measures: The primary outcome is the rate of change in area of GA, based on masked grading by an external Reading Center, of fundus photography in the study eye and fellow eye at two years compared with baseline. Secondary outcomes will include worsening of best-corrected visual acuity (BCVA) of three or more lines (15 or more letters), changes in area of GA as measured on autofluorescence, changes in drusen volume as measured by optical coherence tomography, changes in photoreceptor outer segment (PROS) thickness as measured by optical coherence tomography, as well as changes in drusen area based on masked digital grading of fundus photographs. Safety outcomes will include the number and severity of systemic and ocular toxicities, adverse events and infections.

ELIGIBILITY:
Inclusion Criteria

1. Participant must be older than 55 years of age.
2. Participant must understand and sign the protocol's informed consent document.
3. Participant must have at least ½ disc area (approximately 1 mm^2) of GA compatible with AMD present in each eye. GA is defined as one or more well-defined, usually more or less circular patches of partial or complete de-pigmentation of the RPE, typically with exposure of underlying choroidal blood vessels. Even if much of the RPE appears to be preserved and large choroidal vessels are not visible, a round patch of RPE partial de-pigmentation may still be classified as early GA. The GA in each eye must be able to be photographed in their entirety.
4. Participant must have at least one large druse (more than or equal to 125 μm) in each eye.
5. Participant must have a steady fixation in both eyes in the foveal or parafoveal area and media clear enough for good quality photographs. This will permit randomization.
6. Participant must have visual acuity between 20/20 and 20/400 in each eye.
7. Female participants must be considered post-menopausal and must not be breast-feeding. Female participants over age 55 who have not had a period for one year will be considered post-menopausal.

Exclusion Criteria

1. Participant is in another investigational study and actively receiving study therapy.
2. Participant is unable to comply with study procedures or follow-up visits.
3. Participant has evidence of ocular disease other than AMD in either eye that may confound the outcome of the study (e.g., diabetic retinopathy with 10 or more hemorrhages or microaneurysms, uveitis, pseudovitelliform macular degeneration moderate/severe myopia).
4. Participant has any of the following: a) a history of macular laser, b) a history of photodynamic therapy (PDT), c) received an intravitreal injection of anti-vascular endothelial growth factor (VEGF) agent for wet/exudative AMD at any point, d) received an intravitreal injection of any other agent (not an anti-VEGF agent) within four months prior to study enrollment or e) received topical treatment of any agent for advanced AMD within one month prior to enrollment. Participants currently taking or who have previously taken AREDS vitamin supplementation are not excluded.
5. Participant has had a vitrectomy.
6. Participant is expected to need ocular surgery during the course of the trial.
7. Participant has undergone lens removal in the last three months or yttrium aluminum garnet (YAG) laser capsulotomy within the last month.
8. Participant is on chemotherapy.
9. Participant is on immunosuppressive medication.
10. Participant is on ocular or systemic medications known to be toxic to the lens, retina or optic nerve.
11. Participant with a history of ocular herpes simplex virus (HSV).
12. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control).
13. History of cancer (other than a non-melanoma skin cancer) diagnosed within the past five years.
14. Laboratory values outside normal limits and considered clinically significant by the investigator.
15. Participant is currently taking one of the following drugs: amprenavir, atazanavir, clarithromycin, darunavir, delavirdine, erythromycin, fluconazole (at doses of 200 mg or greater), fluvoxamine, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, posaconazole, quinupristin, ritonavir, saquinavir, telithromycin, troleandomycin, verapamil or voriconazole.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-10; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wai T. Wong, MD, PhD, Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Klein R, Klein BE, Jensen SC, Meuer SM. The five-year incidence and progression of age-related maculopathy: the Beaver Dam Eye Study. Ophthalmology. 1997 Jan;104(1):7-21. doi: 10.1016/s0161-6420(97)30368-6. PMID 9022098
- [Background] Klein R, Klein BE, Linton KL. Prevalence of age-related maculopathy. The Beaver Dam Eye Study. Ophthalmology. 1992 Jun;99(6):933-43. doi: 10.1016/s0161-6420(92)31871-8. PMID 1630784
- [Background] Seddon JM, Ajani UA, Sperduto RD, Hiller R, Blair N, Burton TC, Farber MD, Gragoudas ES, Haller J, Miller DT, et al. Dietary carotenoids, vitamins A, C, and E, and advanced age-related macular degeneration. Eye Disease Case-Control Study Group. JAMA. 1994 Nov 9;272(18):1413-20. PMID 7933422
- [Result] Wong WT, Dresner S, Forooghian F, Glaser T, Doss L, Zhou M, Cunningham D, Shimel K, Harrington M, Hammel K, Cukras CA, Ferris FL, Chew EY. Treatment of geographic atrophy with subconjunctival sirolimus: results of a phase I/II clinical trial. Invest Ophthalmol Vis Sci. 2013 Apr 26;54(4):2941-50. doi: 10.1167/iovs.13-11650. PMID 23548622

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sirolimus
Started | 11
Completed | 1
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Sirolimus
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.4 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Rate of Change in Area of Geographic Atrophy (GA) in the Study Eye at 24 Months as Compared to Baseline
Description: One Macular Photocoagulation Study Disc Area (MPS DA) is equivalent to 1.77 mm^2 on the retina.
Time Frame: Baseline and Month 24
Measure: Mean (Standard Deviation); unit: MPS DA/month
Arm/Group | Sirolimus
Number analyzed (Participants) | 8
MPS DA/month | 0.102 (0.049)

2. Primary Outcome: Rate of Change in Area of Geographic Atrophy (GA) in the Fellow Eye at 24 Months as Compared to Baseline
Description: One Macular Photocoagulation Study Disc Area (MPS DA) is equivalent to 1.77 mm^2 on the retina.
Time Frame: Baseline and Month 24
Measure: Mean (Standard Deviation); unit: MPS DA/month
Arm/Group | Sirolimus
Number analyzed (Participants) | 8
MPS DA/month | 0.087 (0.034)

3. Secondary Outcome: Number of Study Eyes With a 15 Letter Drop From Baseline at 24 Months
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
Time Frame: Baseline and Month 24
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 8
Number analyzed (Eyes) | 8
eyes | 4

4. Secondary Outcome: Absolute Change in Total Area of Geographic Atrophy (GA) in the Study Eye at 24 Months as Compared to Baseline
Description: Geographic atrophy (GA) is the death of photoreceptors and surrounding cells in the retina. The death of these photoreceptors results in lesions that cause vision loss. The area of GA was determined using planimetry for color stereoscopic fundus images by masked graders at the Doheny Image Reading Center (University of Southern California, Los Angeles, CA).
  This outcome measure was calculated by subtracting the GA value for the study eye at baseline from the GA value for the study eye at Month 24.
  One Macular Photocoagulation Study Disc Area (MPS DA) is equivalent to 1.77 mm^2 on the retina.
Time Frame: Baseline and Month 24
Measure: Mean (Standard Deviation); unit: MPS DA
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 8
Number analyzed (Eyes) | 8
MPS DA | 2.46 (1.18)

5. Secondary Outcome: Absolute Change in Total Area of Geographic Atrophy (GA) in the Fellow Eye at 24 Months as Compared to Baseline
Description: Geographic atrophy (GA) is the death of photoreceptors and surrounding cells in the retina. The death of these photoreceptors results in lesions that cause vision loss. The area of GA was determined using planimetry for color stereoscopic fundus images by masked graders at the Doheny Image Reading Center (University of Southern California, Los Angeles, CA).
  This outcome measure was calculated by subtracting the GA value for the fellow eye at baseline from the GA value for the study eye at Month 24.
  One Macular Photocoagulation Study Disc Area (MPS DA) is equivalent to 1.77 mm^2 on the retina.
Time Frame: Baseline and Month 24
Measure: Mean (Standard Deviation); unit: MPS DA
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 8
Number analyzed (Eyes) | 8
MPS DA | 2.08 (0.83)

6. Secondary Outcome: Relative Change in Total Area of Geographic Atrophy (GA) in the Study Eye at 24 Months as Compared to Baseline
Description: Geographic atrophy (GA) is the death of photoreceptors and surrounding cells in the retina. The death of these photoreceptors results in lesions that cause vision loss. The area of GA was determined using planimetry for color stereoscopic fundus images by masked graders at the Doheny Image Reading Center (University of Southern California, Los Angeles, CA).
  This outcome measure was calculated by dividing the absolute change in the total area of GA in the study eye at 24 months by the baseline value.
  One Macular Photocoagulation Study Disc Area (MPS DA) is equivalent to 1.77 mm^2 on the retina. As the unit of measure for both the absolute change in the total area of GA and the baseline value for the total area of GA is MPS DA, the unit of measure for the relative change in the total area of GA is "ratio."
Time Frame: Baseline to Month 24
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 8
Number analyzed (Eyes) | 8
Ratio | 0.55 (0.62)

7. Secondary Outcome: Relative Change in Total Area of Geographic Atrophy (GA) in the Fellow Eye at 24 Months as Compared to Baseline
Description: Geographic atrophy (GA) is the death of photoreceptors and surrounding cells in the retina. The death of these photoreceptors results in lesions that cause vision loss. The area of GA was determined using planimetry for color stereoscopic fundus images by masked graders at the Doheny Image Reading Center (University of Southern California, Los Angeles, CA).
  This outcome measure was calculated by dividing the absolute change in the total area of GA in the fellow eye at 24 months by the baseline value.
  One Macular Photocoagulation Study Disc Area (MPS DA) is equivalent to 1.77 mm^2 on the retina. As the unit of measure for both the absolute change in the total area of GA and the baseline value for the total area of GA is MPS DA, the unit of measure for the relative change in the total area of GA is "ratio."
Time Frame: Baseline and Month 24
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 8
Number analyzed (Eyes) | 8
Ratio | 0.40 (0.25)

8. Secondary Outcome: Change in Total Area of Drusen in the Study Eye at 24 Months as Compared to Baseline
Description: The total area occupied by drusen was determined using planimetry for color stereoscopic fundus images by masked graders at the Doheny Image Reading Center (University of Southern California, Los Angeles, CA).
  One Macular Photocoagulation Study Disc Area (MPS DA) is equivalent to 1.77 mm^2 on the retina.
Time Frame: Baseline and Month 24
Measure: Mean (Standard Deviation); unit: MPS DA
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 8
Number analyzed (Eyes) | 8
MPS DA | 0.04 (0.58)

9. Secondary Outcome: Change in Total Area of Drusen in the Fellow Eye at 24 Months as Compared to Baseline
Description: as for outcome 8
Time Frame: Baseline and Month 24
Measure: Mean (Standard Deviation); unit: MPS DA
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 8
Number analyzed (Eyes) | 8
MPS DA | 0.08 (0.36)

10. Secondary Outcome: Change in Drusen Volume as Measured by Optical Coherence Tomography (OCT) at 24 Months as Compared to Baseline
Time Frame: Baseline and Month 24
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Sirolimus
Number analyzed (Participants) | 8
mm^3 | 0.04 (0.58)

11. Secondary Outcome: Change in Photoreceptor Outer Segment (PROS) Thickness as Measured by Optical Coherence Tomography at 24 Months as Compared to Baseline
Time Frame: Baseline and Month 24
Population: The PROS thickness analysis was not performed. As a result, data were not collected for this outcome measure.
Arm/Group | Sirolimus
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 42 months
Arm/Group | Sirolimus
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=11)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=11)
Eye discharge (Eye disorders) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1)
Eye irritation (Eye disorders) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood chloride increased (Investigations) | 1 (1)
Blood creatine phosphokinase decreased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Blood magnesium increased (Investigations) | 4 (4)
Blood phosphorus decreased (Investigations) | 1 (1)
Blood potassium increased (Investigations) | 2 (2)
Blood uric acid increased (Investigations) | 1 (1)
Blood urine (Investigations) | 1 (1)
Carbon dioxide increased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2)
Haemoglobin increased (Investigations) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (2)
Lymphocyte count decreased (Investigations) | 1 (1)
Mean cell volume increased (Investigations) | 1 (1)
Monocyte count increased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 2 (2)
Protein total decreased (Investigations) | 1 (1)
Red blood cell count decreased (Investigations) | 1 (1)
Red blood cells urine positive (Investigations) | 2 (2)
Red cell distribution width increased (Investigations) | 1 (1)
Urine ketone body present (Investigations) | 1 (1)
Urine leukocyte esterase (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 2 (2)
White blood cells urine (Investigations) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4)
Headache (Nervous system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Cataract operation (Surgical and medical procedures) | 1 (2)
Varicose vein (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No